CLINICAL TRIAL: NCT05839184
Title: The Effectiveness of the Therapeutic Toys on the Comfort Level of the Infants During Intravenous Canula Insertion
Brief Title: The Effectiveness of the Therapeutic Toys During Intravenous Canula Insertion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Collaborators: Izmir Can Hospital (Unknown)
Responsible Party: Principal Investigator, ESRA ARDAHAN AKGUL, Assistant Professor, Principal Investigator, Izmir Katip Celebi University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 132
Record Dates: First submitted 2023-04-18; First posted 2023-05-03 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Pain, Acute; Comfort
Keywords: pain, comfort
MeSH Terms: conditions — Acute Pain; Pain

STUDY DESIGN:
Intervention Model Description: randomised controlled
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CONTROL GROUP (No Intervention): All newborns in the study will be monitored during IV catheter placement. Newborns in the control group will not be given any therapeutic toy and IV catheter will be placed and their comfort levels and vital signs will be monitored.
- therapeutic toy GROUP (Active Comparator): All newborns in the study will be monitored during IV catheter placement. Newborns in the therapeutic toy group will be given an octopus-shaped therapeutic toy that they can hold in their hands throughout the procedure and IV catheter will be inserted and their comfort levels and vital signs will be monitored.
  Interventions: Device: therapeutic toy

INTERVENTIONS:
Device: therapeutic toy — Neonates in the therapeutic toy group will be given an octopus-shaped therapeutic toy that they can hold in their hands throughout the procedure and IV catheter will be inserted and their comfort levels and vital signs will be monitored.
  Arms: therapeutic toy GROUP

SUMMARY:
Pain relief interventions in invasive interventions are divided into two pharmacologic methods and non-pharmacologic methods. Nonpharmacologic interventions are an area where nurses can easily demonstrate their independent roles. Especially today, when the use of complementary and alternative medicine (CAM) methods is increasing, nurses are also turning to these methods.

Non-pharmacological methods include listening to white noise, non-nutritive sucking, aromatherapy applications, placing the baby on the mother's lap, changing position, rocking, touching, distracting, listening to music, watching cartoons, singing, breastfeeding and giving sucrose solution with breast milk, giving toys and smelling mother odour.

This study was planned to determine the effect of the therapeutic toy used during IV catheter placement, which is the most common invasive intervention in the Neonatal Care Unit where a newborn baby is hospitalized, on the comfort level, crying time and physiological parameters of the newborn.

DETAILED DESCRIPTION:
Comfort is defined as "the expected result with a complex structure within biopsychosocial and environmental integrity in order to provide help, peace of mind and cope with problems related to one's needs". According to Kolcaba, comfort is the experience of relief, peace of mind and meeting needs to solve problems. The term comfort has been frequently used in recent years for infants receiving health care in Neonatal and Neonatal Surgery Intensive Care Units. Physical characteristics of the clinic, immaturity of newborns, frequent routine care and invasive procedures (burn dressing, hydrotherapy, blood collection, IV catheter insertion, heel prick, aspiration, nasogastric catheter insertion, foley catheter insertion, rectal tube insertion, neonatal eye examination) cause a decrease in the comfort of newborns.

As a result of rapidly increasing technological developments, changes are also seen in the neonatal discipline and perinatal mortality rates are decreasing, especially in developing countries. As a result of this development, survival rates of very low birth weight newborns have increased to 85%. Although mortality has decreased in preterm infants, neurodevelopmental, pulmonary and cardiac problems have increased. When the causes of neurodevelopmental problems in preterm infants are examined, it is seen that in addition to retinopathy, systemic infections, nutritional problems due to necrotizing enterocolitis and similar causes, intracranial haemorrhage, there are also stressors such as invasive procedures, pain, noise and light that the newborn is exposed to in the intensive care unit. Stress has negative effects on neurodevelopment.

Newborns who have not reached neurodevelopmental maturity begin to experience stress when they leave their warm, dark, quiet and calm environments that contribute to their brain development and start to receive health care in intensive care units where they are exposed to noisy, light and painful procedures. This stress and invasive sensory experiences are thought to suppress the development of cell migration, synaptogenesis, myelinization and organizational structures in the infant's nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Parent's approval to participate in the study
* Born older than 24th gestational week
* The baby is hospitalized in the Neonatal Intensive Care Clinic
* Need for opening an IV catheter
* A saturation value above 90% before the invasive procedure
* Heart rate between 120-160 beats/min before the invasive procedure
* Respiratory rate between 30-60 breaths/min before invasive procedure
* Ability to open an IV road on the first attempt

Exclusion Criteria:

* The parent is not willing to participate in the study
* The baby is taking any medication that affects the comfort level
* Being monitored with mechanical ventilation
* Failure to open an IV road on the first attempt

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2023-04-20 (Actual); Primary Completion 2023-05-10 (Actual); Study Completion 2023-05-13 (Actual)

PRIMARY OUTCOMES:
COMFORT LEVEL | immediately after the IV catheter insertion,
  The Neonatal Comfort Scale was developed by Ambuel et al., revised by van Dijk et al. and validated in Turkish by Kahraman et al. in 2014. The scores that can be obtained from the Neonatal Comfort Behavior Scale vary between 6-30. A higher score means that the newborn is not comfortable and needs interventions to provide comfort.
COMFORT LEVEL | 1st minute after the IV catheter insertion
  The Neonatal Comfort Scale was developed by Ambuel et al., revised by van Dijk et al. and validated in Turkish by Kahraman et al. in 2014. The scores that can be obtained from the Neonatal Comfort Behavior Scale vary between 6-30. A higher score means that the newborn is not comfortable and needs interventions to provide comfort.
COMFORT LEVEL | 5th minute after the IV catheter insertion
  The Neonatal Comfort Scale was developed by Ambuel et al., revised by van Dijk et al. and validated in Turkish by Kahraman et al. in 2014. The scores that can be obtained from the Neonatal Comfort Behavior Scale vary between 6-30. A higher score means that the newborn is not comfortable and needs interventions to provide comfort.
BREATHE PER MINUTE | immediately after the IV catheter insertion
  The form was created by the researchers by reviewing the literature in order to collect physiological parameter data just before the intervention was applied to the newborn, when the intervention started and 1 minute and 5 minutes after the intervention ended.
BREATHE PER MINUTE | 1st minute after the IV catheter insertion
  The form was created by the researchers by reviewing the literature in order to collect physiological parameter data just before the intervention was applied to the newborn, when the intervention started and 1 minute and 5 minutes after the intervention ended.
BREATHE PER MINUTE | 5th minute after the IV catheter insertion
  The form was created by the researchers by reviewing the literature in order to collect physiological parameter data just before the intervention was applied to the newborn, when the intervention started and 1 minute and 5 minutes after the intervention ended.
HEARTH RATE PER MINUTE | immediately after the IV catheter insertion
  The form was created by the researchers by reviewing the literature in order to collect physiological parameter data just before the intervention was applied to the newborn, when the intervention started and 1 minute and 5 minutes after the intervention ended.
HEARTH RATE PER MINUTE | 1st minute after the IV catheter insertion
  The form was created by the researchers by reviewing the literature in order to collect physiological parameter data just before the intervention was applied to the newborn, when the intervention started and 1 minute and 5 minutes after the intervention ended.
HEARTH RATE PER MINUTE | 5th minute after the IV catheter insertion
  The form was created by the researchers by reviewing the literature in order to collect physiological parameter data just before the intervention was applied to the newborn, when the intervention started and 1 minute and 5 minutes after the intervention ended.
OXYGEN SATURATION | immediately after the IV catheter insertion
  The form was created by the researchers by reviewing the literature in order to collect physiological parameter data just before the intervention was applied to the newborn, when the intervention started and 1 minute and 5 minutes after the intervention ended.
OXYGEN SATURATION | 1st minute after the IV catheter insertion
  The form was created by the researchers by reviewing the literature in order to collect physiological parameter data just before the intervention was applied to the newborn, when the intervention started and 1 minute and 5 minutes after the intervention ended.
OXYGEN SATURATION | 5th minute after the IV catheter insertion
  The form was created by the researchers by reviewing the literature in order to collect physiological parameter data just before the intervention was applied to the newborn, when the intervention started and 1 minute and 5 minutes after the intervention ended.

SECONDARY OUTCOMES:
DURATION OF CRYING | Procedure (During the IV catheter insertion process)
  During the IV catheter insertion process, the time will be measured with a stopwatch from the first moment the baby cries until the last moment.

CONTACTS AND LOCATIONS:
Overall Officials: Esra ARDAHAN AKGÜL, Asst. Prof., Study Chair — İzmir Katip Çelebi University
Locations (1):
- Katip Celebi University, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No